CLINICAL TRIAL: NCT03644992
Title: An Analysis Into the Cause and Preventional Method of Thromboembolic Disease in Gynecological Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2018-07-232
Record Dates: First submitted 2018-08-21; First posted 2018-08-24 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Thromboembolic Disease; Gynecological Surgery
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thromboembolic Disease: the patients who undergo gynecological operations but develop thromboembolic disease

SUMMARY:
The aim of this cross-sectional study is to describe the specific situations of thromboembolic disease in gynecological surgery and identify the risk factors of it.

DETAILED DESCRIPTION:
The electronic medical data of 54 patients who undergo operations to treat gynecological diseases but develop thromboembolic disease will be analyzed retrospectively in this study. The location, symptom and other situations of embolism will be described and multiple linear analyse will be employed to identify the risk factors of it.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study with informed consent;
2. Females aged 20-80 who are confirmed with some gynecological diseases and are treated with surgery but embolism happens unfortunately.

Exclusion Criteria:

1. Pregnancy, lactation, postmenopause, or planned pregnancy within two years;
2. Patients with blood diseases prone to thrombosis and those with a history of thrombus were excluded;
3. History of hyperparathyroidism, infectious diseases (tuberculosis, AIDS), autoimmune diseases, or digestive system diseases (malabsorption, crohn disease and dysentery);
4. Other diseases or heavy injuries that will interfere with the results;
5. Simultaneous participation in another clinical study with investigational medicinal product(s) or researcher thinks the subjects are not suitable for this trial.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned sample size was based on data from a previous study, in which the standard deviation was 5. We assumed an one-tailed α error of 0.05 and a sampling error of 1.0. we propose to enroll 60 participants and allow for a dropout rate of 10% for an effective sample size of 54.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
the percentage of different symptoms of thromboembolic disease(%) | 10 months after the operation
  different patients will have various symptoms of embolism like dyspnea, chest pain, hemoptysis and syncope. And we plan to describe the distribution of it.

SECONDARY OUTCOMES:
the location of embolism | 10 months after the operation
  embolism can occur in different parts like the brain, limb, pulmonary and coronary systems. We plan to summarize the location of embolism.
the risk factors of thromboembolic disease | 10 months after the operation
  Performing multiple linear regression analysis with statistical product and service solutions(SPSS) 17.0, we plan to identify the risk factors which can increase the possibility of thromboembolic disease from possible factors like hypertension, diabetes, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- TING LI, Wenzhou, Zhejiang, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03644992/Prot_SAP_000.pdf